CLINICAL TRIAL: NCT05905549
Title: Extended Pancreatic Transection Versus Conventional Pancreatic Transection During Laparoscopic Pancreaticoduodenectomy: a Retrospective Propensity Score-matched Comparison
Brief Title: Extended Pancreatic Transection Versus Conventional Pancreatic Transection During Laparoscopic Pancreaticoduodenectomy
Status: Unknown | Type: Observational
Last Known Status: Not yet recruiting
Sponsor: Xinrui Zhu，MD (Other)
Responsible Party: Sponsor-Investigator, Xinrui Zhu，MD, attending doctor, West China Hospital
Organization: West China Hospital (Other)
Other Study IDs: 2023-167-2
Record Dates: First submitted 2023-06-05; First posted 2023-06-15 (Actual); Last update posted 2023-07-18 (Actual); Status verified 2023-07

CONDITIONS: Laparoscopic Pancreaticoduodenectomy
Keywords: laparoscopic pancreaticoduodenectomy; pancreatic transection level

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- extended pancreatic transection cohort: cases in which the pancreatic transection was performed at the pancreatic neck beyond the left side of the mesenterico-portal axis during laparoscopic pancreaticoduodenectomy, as judged by postoperative abdominal CT scan.
  Interventions: Procedure: extended pancreatic transection during laparoscopic pancreaticoduodenectomy
- conventional pancreatic transection cohort: cases in which the pancreatic transection was performed at the pancreatic neck above the mesenterico-portal axis during laparoscopic pancreaticoduodenectomy, as judged by postoperative abdominal CT scan.

INTERVENTIONS:
Procedure: extended pancreatic transection during laparoscopic pancreaticoduodenectomy — the pancreatic transection was performed at the pancreatic neck beyond the left side of the mesenterico-portal axis during laparoscopic pancreaticoduodenectomy
  Groups: extended pancreatic transection cohort

SUMMARY:
The level of pancreatic neck transection during laparoscopic pancreaticoduodenectomy (LPD) is not conclusive. Theoretically, the level of pancreatic transection can significantly affect the occurrence of postoperative pancreatic fistula (POPF) by influencing both the blood supply to the anastomosis and the location of the main pancreatic duct in the pancreatic transverse section. The investigators conduct a retropective propensity score-matched comparison to compare the impact of extended pancreatic transection and conventional pancreatic transection on POPF and the performance of the pancreaticojejunostomy during LPD.

ELIGIBILITY:
Inclusion Criteria:

1. consecutive patients underwent elective laparoscopic pancreaticoduodenectomy within October 2019 to April 2023
2. the perioperative and follow-up study data information can be collected completely
3. The level of pancreatic neck dissection can be determined by postoperative abdominal CT
4. patients without the history of neoadjuvant chemotherapy or radiotherapy

Exclusion Criteria:

1. conversion to laparotomy due to various reasons during operation;
2. combined with resection and reconstruction of the portal vein or the superior mesenteric vein
3. combined with other organ resection
4. the perioperative and follow-up study data information can not be collected completely, or the level of pancreatic neck dissection can not be determined by postoperative abdominal CT
5. patients with the history of neoadjuvant chemotherapy or radiotherapy
6. the main pancreatic duct did not be found during the operation, the duct-to-mucosa pancreaticojejunostomy could not be performed

Ages: 18 Years to 90 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: patients who had underwent laparoscopic pancreaticoduodenectomy
Sampling Method: Non-Probability Sample
Enrollment: 184 (Estimated)
Dates: Start 2023-08-01 (Estimated); Primary Completion 2023-12-30 (Estimated); Study Completion 2024-06-30 (Estimated)

PRIMARY OUTCOMES:
the incidence of clinically relevant pancreatic fistula | 3 months postoperatively
  the incidence of the clinically relevant pancreatic fistula according the International Study Group of Pancreatic Surgery's definition and grading

SECONDARY OUTCOMES:
surgical performance of pancreaticojejunostomy | intraoperatively
  the duration of pancreaticojejunostomy
postoperative morbidity | 3 months postoperatively
  postoperative morbidity (Clavien-Dindo score ≥3) within 3 months postoperatively
postoperative mortality | 3 months postoperatively
  mortality within 3 months postoperatively

CONTACTS AND LOCATIONS:
Overall Officials: Bing Peng, Study Chair — West China Hospital

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Bardol T, Delicque J, Hermida M, Herrero A, Guiu B, Fabre JM, Souche R. Neck transection level and postoperative pancreatic fistula after pancreaticoduodenectomy: A retrospective cohort study of 195 patients. Int J Surg. 2020 Oct;82:43-50. doi: 10.1016/j.ijsu.2020.08.001. Epub 2020 Aug 22. PMID 32841726
- [Background] Jwa EK, Hwang S. Extended pancreatic transection for secure pancreatic reconstruction during pancreaticoduodenectomy. Ann Hepatobiliary Pancreat Surg. 2017 Aug;21(3):138-145. doi: 10.14701/ahbps.2017.21.3.138. Epub 2017 Aug 31. PMID 28990000
- [Background] Strasberg SM, Drebin JA, Mokadam NA, Green DW, Jones KL, Ehlers JP, Linehan D. Prospective trial of a blood supply-based technique of pancreaticojejunostomy: effect on anastomotic failure in the Whipple procedure. J Am Coll Surg. 2002 Jun;194(6):746-58; discussion 759-60. doi: 10.1016/s1072-7515(02)01202-4. PMID 12081065